CLINICAL TRIAL: NCT00507559
Title: The Pivotal Study of the Aptus Endovascular AAA Repair System
Acronym: STAPLE-2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiovascular (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2007-01
Record Dates: First submitted 2007-07-24; First posted 2007-07-26 (Estimated); Results first posted 2016-05-27 (Estimated); Last update posted 2021-11-03 (Actual); Status verified 2021-10

CONDITIONS: Abdominal Aortic Aneurysms (AAA)
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- AAA Repair System (Experimental)
  Interventions: Device: Aptus Endovascular AAA Repair System

INTERVENTIONS:
Device: Aptus Endovascular AAA Repair System — EVAR (endovascular aneurysm repair)

SUMMARY:
A prospective, non-randomized, multi-center clinical study to evaluate the safety and effectiveness of the Aptus Endovascular AAA Repair System compared to an open surgical repair historical control group in the treatment of abdominal aortic aneurysms (AAA).

DETAILED DESCRIPTION:
The historical group is the open surgical repair procedures (n=323) in the Lifeline Foundation (now American Vascular Association Foundation).

ELIGIBILITY:
Inclusion Criteria:

* Infrarenal AAA with a maximum diameter ≥ 4.5 cm.
* Infrarenal AAA with at least 12 mm length of non-aneurysmal proximal neck.
* Infrarenal AAA with a proximal neck internal diameter between 19-29 mm.
* Infrarenal AAA with an internal diameter at the aortic bifurcation ≥ 18 mm.
* Infrarenal AAA with an angle of ≤ 60° relative to the long axis of the aneurysm.
* Bilateral iliac artery distal fixation sites ≥ 10 mm in length.
* Bilateral iliac arteries with an internal diameter between 9 and 20 mm.
* Bilateral femoral/iliac arteries with morphology compatible with standard vascular access techniques and vessel size must accommodate a 16F (5.3 mm) or 18F (6.0 mm) delivery system.

Exclusion Criteria:

* Myocardial infarction within past 10 weeks.
* Active systemic infection.
* Ruptured or leaking AAA.
* Mycotic or inflammatory AAA.
* Genetic connective tissue disorders (e.g., Marfans or Ehlers-Danlos Syndromes).
* Concomitant TAA or thoracoabdominal aortic aneurysms.
* Requires emergent AAA surgery.
* Previous AAA repair.
* Patients with a body habitus that would prevent imaging required by the study.
* Patient has significant comorbid conditions that pose undue risk of general anesthesia or endovascular surgery.
* Patient requires additional planned major procedure at the time of AAA repair or within 30 days before or after AAA repair.
* Dialysis dependent renal failure or creatinine > 2.5 mg/dL.
* Allergy to or intolerance of radiopaque contrast agents.
* Patients with a known sensitivity or allergy to implant materials.
* Patients who cannot discontinue oral anticoagulation or antiplatelet therapy at the time of the study procedure.
* Patients with history of bleeding diathesis or hypercoagulable condition.
* Patients with thrombus, calcification, and/or plaque ≥ 2mm in thickness and/or ≥ 50% (180°) continuous coverage of the vessel circumference in the intended seal zone.
* Patients with irregular shaped calcification and/or plaque that may compromise the fixation and sealing at the proximal or distal implantation sites.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2007-09; Primary Completion 2010-03 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald M Fairman, M.D, Principal Investigator — University of Pennsylvania; Manish Mehta, M.D, Principal Investigator — Albany Medical College & Albany Medical Center
Locations (2):
- United States (2):
  - The Vascular Group, Albany, New York
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Groups:
- AAA Repair System: Aptus Endovascular AAA Repair System: EVAR
Period: Overall Study
Arm/Group | AAA Repair System
Started | 155
Completed | 84
Not Completed | 71

BASELINE CHARACTERISTICS:
Arm/Group | AAA Repair System
Number analyzed (Participants) | 155
Age, Continuous [Mean (Standard Deviation); unit: years] | 73 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 145
Region of Enrollment [Number; unit: participants]
  United States | 155

OUTCOME MEASURES:

1. Primary Outcome: Effectiveness: Composite Success Rate
Description: Composite endpoint of delivery success, absence of Type I/III endoleak requiring intervention post-index procedure, absence of migration (>10mm), and absence of aneurysm rupture or conversion.This composite endpoint is compared to an estimated success rate of 80%.
Time Frame: 12 months
Measure: Number; unit: participants
Arm/Group | AAA Repair System
Number analyzed (Participants) | 155
participants | 4

2. Primary Outcome: Safety: MAE (Major Adverse Event)
Description: Percentage (number) of subjects experiencing one or more of major adverse events within the first 30 days post-index procedure compared to the open surgical repair historical group
Time Frame: 30 days
Measure: Number; unit: participants
Arm/Group | AAA Repair System
Number analyzed (Participants) | 155
participants | 3
Statistical Analysis 1: Comparison: AAA Repair System; This is compared to a historical control group, in which 11.1% of subjects experienced one or more MAE within 30 days; Test type: Superiority or Other; p < 0.001, Fisher Exact

3. Secondary Outcome: Safety: SAE (Serious Adverse Event)
Description: Percent (number) of subjects experiencing one or more serious adverse event through 5 years post-index procedure
Time Frame: 5 years
Measure: Number; unit: participants
Arm/Group | AAA Repair System
Number analyzed (Participants) | 155
participants | 129

4. Secondary Outcome: Effectiveness: Surgical Conversion
Description: Percent (number) of subjects undergoing surgical conversion through 12 months post-index procedure.
  Conversion is defined as the patient undergoing open surgical aneurysm repair with partial or complete removal of the study device.
Time Frame: 12 months
Population: 143 reflects the number of subjects with data for the 12 month visit.
Measure: Number; unit: participants
Arm/Group | AAA Repair System
Number analyzed (Participants) | 143
participants | 1

5. Secondary Outcome: Effectiveness: Aneurysm Rupture
Description: Percent (number) of subjects experiencing aneurysm rupture through 12 months post-index procedure
Time Frame: 12 months
Population: 143 reflects the number of subjects with data for the 12 month visit.
Measure: Number; unit: participants
Arm/Group | AAA Repair System
Number analyzed (Participants) | 143
participants | 1

6. Secondary Outcome: Effectiveness: Aneurysm Change
Description: Percent (number) of subjets experiencing aneurysm change (defined as increase in maximum diameter of >5mm) at 12 months post-index procedure
Time Frame: 12 months
Population: Denominator is number of subjects with assessable imaging. Films are not assessable for aneurysm change if the 30-day scan is not available as a baseline.
Measure: Number; unit: participants
Arm/Group | AAA Repair System
Number analyzed (Participants) | 132
participants | 2

7. Secondary Outcome: Effectiveness: EndoStaple Stent/Fracture
Description: Percent (number) of subjects experiencing an EndoStaple stent/fracture at 12 months post-index procedure
Time Frame: 12 months
Population: Denominator is number of subjects with adequate x-ray imaging available at 12 months
Measure: Number; unit: participants
Arm/Group | AAA Repair System
Number analyzed (Participants) | 119
participants | 0

8. Secondary Outcome: Effectiveness: Prosthesis Migration
Description: Percent (number) of subjects experiencing prothesis migration at 12 months post-index procedure
Time Frame: 12 months
Population: The denominator is the number of subjects with adequate CT imaging available at 12 months
Measure: Number; unit: participants
Arm/Group | AAA Repair System
Number analyzed (Participants) | 133
participants | 0

9. Secondary Outcome: Effectiveness: Type I Endoleak and Type III Endoleak
Description: Percent (number) of subjects experiencing type I endoleak (inadequate or ineffective seal of graft) or III endoleak (inadequate seal of graft joints or graft rupture) requiring intervention through 12 months post-index procedure
Time Frame: 12 months
Population: Denominator is the number of subjects with adequate CT imaging available at 12 months
Measure: Number; unit: participants
Arm/Group | AAA Repair System
Number analyzed (Participants) | 132
participants | 2

10. Secondary Outcome: Effectiveness: Thrombosis
Description: Percent (number) of subjects experiencing thrombosis through 5 years post-index procedure
Time Frame: 5 years
Population: Events classified by the clinical events committee as thrombosis in device, embolism, device occlusion, vascular occlusion and thrombosis were included in the number of patients affected
Measure: Number; unit: participants
Arm/Group | AAA Repair System
Number analyzed (Participants) | 155
participants | 64

ADVERSE EVENTS:
Time Frame: 5 years
Arm/Group | AAA Repair System
Serious Adverse Events (participants affected / at risk) | 129/155
Other Adverse Events (participants affected / at risk) | 148/155
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AAA Repair System (N=155)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1)
Angina pectoris (Cardiac disorders) | 9 (10)
Angina unstable (Cardiac disorders) | 1 (1)
Arrhythmia (Cardiac disorders) | 8 (9)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 7 (8)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1)
Coronary artery disease (Cardiac disorders) | 2 (2)
Coronary artery stenosis (Cardiac disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 9 (9)
Syncope (Cardiac disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Aorto-oesophageal fistula (Gastrointestinal disorders) | 1 (1)
Colitis ischaemic (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 7 (7)
Haemorrhoids (Gastrointestinal disorders) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Large intestine polyp (Gastrointestinal disorders) | 1 (1)
Peptic ulcer perforation (Gastrointestinal disorders) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (2)
Asthenia (General disorders) | 1 (1)
Chest pain (General disorders) | 1 (1)
Death (General disorders) | 1 (1)
Device deployment issue (General disorders) | 1 (1)
Device dislocation (General disorders) | 3 (3)
Device malfunction (General disorders) | 1 (1)
Device occlusion (General disorders) | 5 (6)
Hernia (General disorders) | 1 (1)
Hernia obstructive (General disorders) | 1 (1)
Medical device complication (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Stent-graft endoleak (General disorders) | 12 (15)
Thrombosis in device (General disorders) | 24 (36)
Unevaluable event (General disorders) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1)
Bacteraemia (Infections and infestations) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
Clostridial infection (Infections and infestations) | 1 (1)
Diverticulitis (Infections and infestations) | 2 (2)
Encephalitis viral (Infections and infestations) | 1 (1)
Groin abscess (Infections and infestations) | 1 (1)
Incision site cellulitis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 8 (8)
Urinary tract infection (Infections and infestations) | 2 (2)
Urosepsis (Infections and infestations) | 1 (1)
Wound infection (Infections and infestations) | 2 (2)
Hip fracture (Injury, poisoning and procedural complications) | 3 (3)
Multiple fractures (Injury, poisoning and procedural complications) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 2 (2)
Procedural haemorrhage (Injury, poisoning and procedural complications) | 2 (2)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1)
Urinary retention postoperative (Injury, poisoning and procedural complications) | 1 (1)
Vascular graft occlusion (Injury, poisoning and procedural complications) | 3 (7)
Vascular injury (Injury, poisoning and procedural complications) | 2 (2)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1)
Carcinoembryonic antigen increased (Investigations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1)
Hypovolaemia (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Monarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 (1)
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3)
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Kaposi's sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Meningioma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Oropharyngeal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6)
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Small intestine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Carotid artery stenosis (Nervous system disorders) | 2 (2)
Cerebral haemorrhage (Nervous system disorders) | 2 (2)
Cerebrovascular accident (Nervous system disorders) | 4 (5)
Haemorrhage intracranial (Nervous system disorders) | 1 (1)
Hemiparesis (Nervous system disorders) | 1 (1)
Hydrocephalus (Nervous system disorders) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 1 (1)
Multiple sclerosis (Nervous system disorders) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 4 (5)
Confusional state (Psychiatric disorders) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1)
Nephrotic syndrome (Renal and urinary disorders) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 2 (2)
Renal tubular necrosis (Renal and urinary disorders) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 7 (18)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Aortic aneurysm repair (Surgical and medical procedures) | 1 (1)
Hip arthroplasty (Surgical and medical procedures) | 3 (3)
Intervertebral disc operation (Surgical and medical procedures) | 1 (1)
Intestinal resection (Surgical and medical procedures) | 1 (1)
Large intestine operation (Surgical and medical procedures) | 1 (1)
Aneurysm ruptured (Vascular disorders) | 1 (1)
Aortic stenosis (Vascular disorders) | 1 (1)
Arterial stenosis (Vascular disorders) | 1 (1)
Arteriosclerosis (Vascular disorders) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 3 (3)
Embolism (Vascular disorders) | 9 (11)
Embolism venous (Vascular disorders) | 1 (1)
Femoral artery embolism (Vascular disorders) | 1 (1)
Haematoma (Vascular disorders) | 4 (5)
Hypertension (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 4 (5)
Intermittent claudication (Vascular disorders) | 6 (8)
Orthostatic hypotension (Vascular disorders) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 2 (2)
Peripheral artery aneurysm (Vascular disorders) | 1 (1)
Peripheral artery stenosis (Vascular disorders) | 4 (6)
Peripheral artery thrombosis (Vascular disorders) | 2 (3)
Peripheral ischaemia (Vascular disorders) | 21 (25)
Vascular occlusion (Vascular disorders) | 3 (4)
Vascular stenosis (Vascular disorders) | 4 (6)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AAA Repair System (N=155)
Anaemia (Blood and lymphatic system disorders) | 11 (11)
Arrhythmia (Cardiac disorders) | 9 (10)
Oedema peripheral (General disorders) | 11 (12)
Pyrexia (General disorders) | 17 (17)
Stent-graft endoleak (General disorders) | 51 (55)
Thrombosis in device (General disorders) | 10 (15)
Pneumonia (Infections and infestations) | 8 (9)
Urinary tract infection (Infections and infestations) | 9 (11)
Urinary retention (Renal and urinary disorders) | 10 (10)
Hypertension (Vascular disorders) | 15 (16)
Intermittent claudication (Vascular disorders) | 22 (24)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No